CLINICAL TRIAL: NCT05843669
Title: An Open-label, Multicenter, Single-group Study to Evaluate the Effects of Long-term Use of Mucinex® in Patients With Stable Chronic Bronchitis.
Brief Title: A Study to Explore if Long-term Use of Mucinex Can Help With Symptoms in Patients With Stable Chronic Bronchitis.
Acronym: AHR CB
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: American Health Research (Other)
Collaborators: Vitaccess Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5132-02-2023
Record Dates: First submitted 2023-04-06; First posted 2023-05-06 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Chronic Bronchitis
Keywords: Stable chronic bronchitis; Real-world study; Mucinex; Guafenesin
MeSH Terms: conditions — Bronchitis, Chronic | interventions — Acetylcysteine

STUDY DESIGN:
Intervention Model Description: Phase 4 real-world study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- N/A. Only one arm. (Experimental): Single arm. During the 12-week period of receiving treatment, patient participants will take Mucinex® 12h, 2 x 600 mg (1200 mg total) twice daily and complete weekly bespoke surveys and the CASA-Q instrument.
  Interventions: Drug: Guafenesin tablets

INTERVENTIONS:
Drug: Guafenesin tablets — During the 12-week period of receiving treatment, patient participants will take Mucinex® 12h, 2 x 600 mg (1200 mg total) twice daily.
  Other Names: Mucinex®

SUMMARY:
This is an open-label, multicenter, single-group study designed to determine the effectiveness of Mucinex® when used by patients to treat SCB over a 12-week period, following a 2-week run-in period of no treatment (to establish a baseline).

DETAILED DESCRIPTION:
Data will be collected via the Vitaccess Real[TM] platform from adult patients with SCB and HCPs based in the US. During the 12-week period of receiving treatment, patient participants will take Mucinex® 12h, 2 x 600 mg (1200 mg total) twice daily and complete weekly bespoke surveys and the CASA-Q instrument. Patient-reported data will include prior usage of Mucinex®, treatment compliance, treatment satisfaction, and symptoms.

During this same period of time, HCPs will report treatment satisfaction via electronic case report forms (eCRFs), and will also have the ability to spontaneously report any treatment-emergent adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with a diagnosis of SCB at recruitment, male and female, over 40 years of age
* A Pulmonary Function Test with FEV1/FVC less than 0.7 (70%) at the time of enrollment or at least a 10 year history of cigarette abuse.
* Patients who have chronic sputum production 3 months out of the year for 2 consecutive years and a productive cough as part of their symptoms.
* Patients who understand and are able to fill out a questionnaire and ePRO weekly
* Patients who have not used guaifenesin containing products within one month of the time of study enrollment
* Patients with 6 to 12 (ideally 12)-month historical data - retrieved from either electronic medical records (EMR), electronic health records (EHRs), or provided by the patient via interview.

Rescue medicine:

• No rescue medicine will be provided. Information regarding concurrent rescue medications, either OTC or via prescription, will be collected.

Exclusion Criteria:

* Patients who are pregnant or breastfeeding
* Participation in another study involving an investigational product within 30 days of the baseline visit
* Pulmonary diagnosis other than CB, (such as cystic fibrosis, alpha-1 antitrypsin deficiency, bronchiectasis, or pulmonary fibrosis)
* Active lung cancer or history of lung cancer if it has been less than 2 years since lung resection or other treatment including chemotherapy or radiation. If the patient has a history of lung cancer, they must be in remission
* Psychiatric disorder that precludes participation in the study
* History of alcohol and/or drug abuse within one year of study start
* Patients taking intermittent antibiotics and patients taking oral and systemic corticosteroids (e.g., prednisone at a dose of > 10 mg/day).
* Patients on a chronic stable dose of macrolide antibiotics at the start of the study may be included at the discretion of the Principal Investigator.
* Patients who had an acute exacerbation of chronic bronchitis within a period of one month of starting the study that required systematic steroids or antibiotics
* Hypersensitivity to guaifenesin, or any other excipient listed in the product.

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2023-07-17 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-11-13 (Actual)

PRIMARY OUTCOMES:
Describe patient-reported real-world clinical use of Mucinex® (i.e., prior to study start) in patients with SCB. | At baseline (week 0).
  Patient-reported quantitative data via "Prior usage of Mucinex®" bespoke survey. This comprises three questions regarding patients' previous use of Mucinex, the approximate timing of use, and the frequency of use.
Describe change in patient-reported real-world clinical use of Mucinex® (i.e., treatment compliance) in patients with SCB. | Every 1 week during 12 week period of receiving Mucinex® (week 2 to 14).
  Patient-reported quantitative data via "Treatment compliance" bespoke survey.
Describe change in patient-reported real-world clinical use of Mucinex® (i.e., treatment satisfaction) in patients with SCB. | Every 2 weeks during 12 week period of receiving Mucinex® (week 2 to 14).
  Patient-reported quantitative data via "Treatment satisfaction" bespoke survey.
Describe change in patient-reported real-world clinical use of Mucinex® (i.e., symptoms) in patients with SCB. | Every 1 week during 12 week period of receiving Mucinex® (week 2 to 14).
  Patient-reported quantitative data via "Symptoms" bespoke survey.
Describe change in patient-reported real-world clinical use of Mucinex® (i.e., cough and sputum production and its impact) in patients with SCB. | Every 1 week during 12 week period of receiving Mucinex® (week 2 to 14).
  Patient-reported quantitative data via the Cough and Sputum Assessment Questionnaire, CASA-Q (web- and app-based). This is a validated instrument to measure cough and sputum production, and their impact in patients with chronic obstructive pulmonary disease (COPD) and/or chronic bronchitis
Describe change in HCP-reported real-world clinical use of Mucinex® (i.e., treatment-emergent adverse events) in patients with SCB. | As many times as needed during 12 week period of receiving Mucinex® (week 2 to 14).
  HCP-reported quantitative data via electronic case report forms ("Treatment-emergent adverse events" survey).
Describe change in HCP-reported real-world clinical use of Mucinex® (i.e., treatment satisfaction) in patients with SCB. | At final visit (week 14).
  HCP-reported quantitative data via electronic case report forms ("Treatment satisfaction" survey).
Describe change in HCP-reported real-world clinical use of Mucinex® (i.e., energy levels) in patients with SCB. | At week 8, and at final visit (week 14).
  HCP-reported quantitative data via electronic case report forms ("Energy levels" survey).
Describe change in HCP-reported real-world clinical use of Mucinex® (i.e., healthcare resource use) in patients with SCB. | At baseline visit (week 0), at week 8, and at final visit (week 14).
  HCP-reported quantitative data via electronic case report forms ("Healthcare resource use" survey).

SECONDARY OUTCOMES:
Describe the rate of patient-reported chronic bronchitis ePRO improvements while on treatment with Mucinex® compared to patient history or baseline. | At baseline (week 0), and every 1 week during 14 week study period.
  Patient-reported quantitative data via the Cough and Sputum Assessment Questionnaire, CASA-Q (web- and app-based).
Describe the rate of concomitant rescue and/or maintenance inhaler use while on treatment with Mucinex® compared to patient history/baseline established as part of Medication Record Log completed by HCP in the eCRF at baseline visit. | As many times as needed during 12 week period of receiving Mucinex® (week 2 to 14).
  HCP-reported quantitative data via electronic case report forms ("Treatment-emergent adverse events" survey).
Describe the HCP-reported rate of healthcare resource utilization while on treatment with Mucinex® compared to patient history or baseline. | At baseline visit (week 0), at week 8, and at final visit (week 14).
  HCP-reported quantitative data via electronic case report forms ("Healthcare resource use" survey).
Assess HCP-reported treatment satisfaction of patients while on treatment with Mucinex®. | At final visit (week 14).
  HCP-reported quantitative data via electronic case report forms ("Treatment satisfaction" survey).
Assess patient-reported treatment satisfaction while on treatment with Mucinex®. | Every 2 weeks during 12 week period of receiving Mucinex® (week 2 to 14).
  Patient-reported quantitative data via "Treatment satisfaction" bespoke survey.

OTHER OUTCOMES:
Rate of chronic bronchitis exacerbations in patients who use Mucinex® to manage symptoms of SCB. | As many times as needed during 12 week period of receiving Mucinex® (week 2 to 14).
  HCP-reported quantitative data via electronic case report forms ("Treatment-emergent adverse events" survey).
Change in patient-reported health-related quality of life in patients who use Mucinex® to manage symptoms of SCB | At baseline (week 0), and every 1 week during 14 week study period.
  Patient-reported quantitative data via the Cough and Sputum Assessment Questionnaire, CASA-Q (web- and app-based). This is a validated instrument to measure cough and sputum production, and their impact in patients with chronic obstructive pulmonary disease (COPD) and/or chronic bronchitis
Change in HCP-reported health-related quality of life in patients who use Mucinex® to manage symptoms of SCB. | At week 8, and at final visit (week 14).
  HCP-reported quantitative data via electronic case report forms ("Energy levels" survey).

CONTACTS AND LOCATIONS:
Overall Officials: Selwyn Spangenthal, MD, Principal Investigator — American Health Research; Clinical Research of Rock Hill
Locations (2):
- United States (2):
  - American Health Research, Charlotte, North Carolina
  - Clinical Research of Rock Hill, Rock Hill, South Carolina

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.

REFERENCES:
- [Background] Spangenthal S, Divel C, Borecka O, Fellows A, Llewellyn S. The interplay between CASA-Q domains: insights from a real-world study investigating the effects of extended-release guaifenesin in stable chronic bronchitis. Presented at the 10th American Cough Conference (ACC) 2025; Jun 2025; Dulles, VA, US.
- [Background] Divel C, Spangenthal S, Shea T, Borecka O, Llewellyn S, Adeleke M, Patel P. Adjunctive long-term Mucinex® use leading to improvement in stable chronic bronchitis and decreased health care resource utilization - a case report. Am J Respir Crit Care Med 2025;211:A6293. https://doi.org/10.1164/ajrccm.2025.211.Abstracts.A6293
- [Background] Spangenthal S, Llewellyn S, Borecka O, Pollack C, Adeleke M, Kulasekaran A, Birring S, Mazzone S, Shea T. Real world effectiveness of guaifenesin ER in tackling mucus hypersecretion in stable chronic bronchitis. Presented at The Thirteenth London International Cough Symposium; Jul 18-19; London, UK
- [Background] Divel C, Borecka O, Llewellyn S, Spangenthal S. Assessment of stable chronic bronchitis improvement with adjunctive long-term Mucinex® use via the cough and sputum assessment questionnaire (CASA-Q). Presented at The Annual Meeting of the American College of Chest Physicians (CHEST) 2025; Oct 19-22; Chicago, IL, US.
- [Background] Spangenthal S, Divel C, Borecka O, Llewellyn S. Real-world use of Vitaccess Real™ platform to assess quality of life impact with long-term use of Mucinex® in stable chronic bronchitis. Presented at the 32nd International Society of Quality of Life Research (ISOQOL) Annual Conference 2025; Oct 22-25; Milwaukee, WI, US.
- [Background] Spangenthal S, Divel C, Borecka O, Llewellyn S. Adjunctive long-term use of Mucinex® leading to improvement in stable chronic bronchitis and patient's quality of life: A case report. Medical Reports. 2025;14,100384.
- See also: The Thirteenth London International Cough Symposium research poster — https://www.researchgate.net/publication/382744095
- See also: ACC 2025 presentation — https://www.researchgate.net/publication/391522663
- See also: ISOQOL 2025 research poster — https://www.researchgate.net/publication/394966835_Real-world_use_of_Vitaccess_Real_platform_to_assess_quality_of_life_impact_with_long-term_use_of_MucinexR_in_stable_chronic_bronchitis